CLINICAL TRIAL: NCT05988034
Title: A Multiple-dose, Randomized, Double-blind, Placebo-controlled, Active-Comparator, Parallel Study to Investigate the Effect of Avacopan at Therapeutic and Supratherapeutic Doses on the QT/QTc Interval in Healthy Subjects
Brief Title: A Study to Assess the Effect of Avacopan at Therapeutic and Supratherapeutic Doses on the QT/QTc Interval in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CL014_168
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-07

CONDITIONS: Electrocardiography
Keywords: Complement 5a receptor (C5aR); Anti-neutrophil cytoplasmic antibody-associated vasculitis; Complement; Vasculitis
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Vasculitis | interventions — avacopan; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1: Avacopan (Experimental): Participants will be randomized to receive multiple doses of avacopan orally twice daily (BID): 30 mg for 7 days and 100 mg for 7 days, for a total of 14 dosing days, and placebo for moxifloxacin on Days 1 and 15.
  Interventions: Drug: Avacopan; Drug: Placebo for moxifloxacin
- Cohort 2A: Moxifloxacin/Placebo (Active Comparator): Participants will be randomized to receive moxifloxacin 400 mg orally on Day 1, placebo for avacopan BID on Days 1 to 14, and placebo for moxifloxacin on Day 15.
  Interventions: Drug: Moxifloxacin; Drug: Placebo for avacopan; Drug: Placebo for moxifloxacin
- Cohort 2B: Placebo/Moxifloxacin (Active Comparator): Participants will be randomized to receive placebo for moxifloxacin orally on Day 1, placebo for avacopan BID on Days 1 to 14, and moxifloxacin 400 mg orally on Day 15.
  Interventions: Drug: Moxifloxacin; Drug: Placebo for avacopan; Drug: Placebo for moxifloxacin

INTERVENTIONS:
Drug: Avacopan — Administered orally.
  Arms: Cohort 1: Avacopan
Drug: Moxifloxacin — Administered orally.
  Arms: Cohort 2A: Moxifloxacin/Placebo; Cohort 2B: Placebo/Moxifloxacin
Drug: Placebo for avacopan — Administered orally.
  Arms: Cohort 2A: Moxifloxacin/Placebo; Cohort 2B: Placebo/Moxifloxacin
Drug: Placebo for moxifloxacin — Administered orally.

SUMMARY:
The primary objective of this study is to evaluate the effects of therapeutic and supratherapeutic doses of avacopan on the heart rate corrected QT interval, using Fridericia's formula (QTcF).

ELIGIBILITY:
Inclusion Criteria:

* Be able to verbalize understanding of consent form and able to provide written informed consent;
* Healthy male or female: No known history of a clinically significant medical diagnosis in the opinion of the Investigator and is not receiving prescription medication except birth control therapies; this includes but is not limited to no history of heart or lung disease (including latent tuberculosis), high blood pressure, history of any cardiac or endocrine disease (including thyroid disease and diabetes); appendectomy and cholecystectomy are allowed;
* Aged ≥18 and ≤60 years at the time of screening;
* Body mass index ≥18.0 and ≤30.0 kg/m^2, and body weight of ≥50 kg, at screening and Day -2;
* Non- or ex-smoker; an ex-smoker is defined as someone who completely stopped using nicotine products for at least 180 days prior to the first study drug administration;
* A female participant meeting 1 of the following criteria: (1) female participants of child-bearing potential using adequate contraception during and for at least 90 days after any administration of study medication; or (2) physiological postmenopausal status, defined as the following: absence of menses for at least 1 year prior to the first study drug administration (not due to amenorrhea secondary to lactation); and follicle stimulating hormone (FSH) levels ≥40 mIU/mL at screening; or (3) surgical postmenopausal status, defined as the following: bilateral oophorectomy; and absence of menses for at least 90 days prior to the first study drug administration; and FSH levels ≥40 mIU/mL at screening; or (4) surgical sterilization including tubal ligation, salpingectomy and hysterectomy. If the postmenopausal participant has an FSH of <40 mIU/mL, but meets the above criteria in either (1), (2), (3) or (4) (for all aspects other than FSH levels) as well as all the other inclusion criteria, the participant may be included in the study if the estradiol serum level measured at screening is equal to or below 150 pmol/L. If male, non-vasectomized participants with female partners of child-bearing potential must agree to use contraception and agree not to donate sperm during the study period and for 90 days after the last study drug administration;
* Willing to communicate with an investigator and site staff and comply with all study procedures and requirements.

Exclusion Criteria:

* An uninterpretable or abnormal screening electrocardiogram (ECG) indicating a second- or third-degree atrioventricular block, or one or more of the following: QRS interval >110 msec; QTcF >450 msec; PR interval >200 msec; HR <40 bpm; or any rhythm other than sinus rhythm that is interpreted an investigator to be clinically significant;
* History of risk factors for torsades de pointes, including unexplained syncope, known long QT syndrome, heart failure, myocardial infarction, angina, or clinically significant abnormal laboratory assessments including hypokalemia, hypercalcemia, or hypomagnesemia. Participants will also be excluded if there is a family history of long QT syndrome or Brugada syndrome;
* A sustained supine systolic blood pressure >150 mm Hg or <90 mm Hg or a supine diastolic blood pressure >95 mm Hg or <50 mm Hg at screening or on Day -1. Blood pressure may be retested more than once in the supine position. The blood pressure abnormality is considered sustained if either the systolic or the diastolic pressure values are outside the stated limits after 3 assessments and the participant may not be randomized;
* A resting HR of <40 bpm or >100 bpm when vital signs are measured at screening or on Day -1;
* Unstable cardiovascular disease, including recent myocardial infarction or cardiac arrhythmia;
* History of acquired immunodeficiency syndrome or positive test results for human immunodeficiency virus, hepatitis C virus antibody, or hepatitis B surface antigen at screening;
* Positive urine drug or alcohol screen at screening or on Day -2 (admission);
* Clinically significant illness, including viral syndromes within 3 weeks prior to Day 1;
* Women who are pregnant according to a serum pregnancy test (or planning to become pregnant within the next 6 months) or currently breastfeeding, at screening or according to a urine pregnancy test on Day -2 (admission);
* Participation in another investigational drug or device study or treated with an investigational drug within 30 days or 5 half-lives, whichever is longer, prior to Day 1;
* Received avacopan previously;
* Consumed more than 21 units of ethanol per week at any time in the 6 months prior to Day 1 (1 unit of ethanol is equivalent to 8 ounces of beer, 4 ounces of wine, or 1 ounce of spirits) or history of alcoholism and/or drug/chemical abuse within 5 years;
* Use of prescription medications (with the exception of hormone replacement therapy and hormonal birth control), including nonsteroidal anti-inflammatory drugs or sucralfate and medications known to prolong the QT/QTc interval or herbal preparations within 14 days or 5 half-lives (whichever is longer) prior to Day 1, or use of an over-the-counter medication, vitamins, or supplements (including omega-3 fish oils) within 7 days prior to Day 1;
* Use of alcohol-, caffeine-, or xanthine-containing products, Seville oranges (sour), grapefruit, or grapefruit juice, within 72 hours prior to Day 1;
* Strenuous activity (e.g., sports) from 96 hours (4 days) prior to entry into the clinical research unit (on Day -2) and throughout the study (until the final follow-up visit is conducted);
* Donated more than 500 mL of blood or significant blood loss within 60 days prior to signing the informed consent form;
* Any other medical, psychological, or social condition that, in the opinion of an investigator, would prevent the participant from fully participating in the study, would represent a concern for study compliance, or would constitute a safety concern to the participant;
* An employee of an investigator or study center with direct involvement in the proposed study or other studies under the direction of that investigator or study center, as well as a family member of the employee or investigator;
* Known hypersensitivity to drugs including moxifloxacin;
* Participants taking strong CYP3A4 inducers (e.g., phenytoin, fosphenytoin, rifampicin, carbamazepine, St. John's Wort, nevirapine, pentobarbital, primidone, rifapentine, enzalutamide, lumacaftor, mitotane, apalutamide, quinine, rimexolone, rifaximin, rifamycin, topiramate, oxcarbazepine) or moderate CYP3A4 inducers (e.g., bosentan, efavirenz, etravirine, modafinil, dexamethasone, etravirine, nafcillin, dabrafenib, methotrexate, bexarotene, mifepristone) within 2 weeks prior to prior to Day 1;
* Positive screening tuberculosis blood test.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2019-11-08 (Actual); Primary Completion 2020-01-22 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in QTcF | Day -1 (baseline) and up to Day 14

SECONDARY OUTCOMES:
Change from Baseline in Heart Rate (HR) | Day -1 (baseline) and Days 1, 7, and 14
Change from Baseline in Time Between P and R Wave (PR Interval) | Day -1 (baseline) and Days 1, 7, and 14
Change from Baseline in Complex Between Q and S Wave (QRS Interval) | Day -1 (baseline) and Days 1, 7, and 14
Placebo-corrected Change from Baseline in HR | Day -1 (baseline) and Days 1, 7, and 14
Placebo-corrected Change from Baseline in QTcF | Day -1 (baseline) and Days 1, 7, and 14
Placebo-corrected Change from Baseline in PR Interval | Day -1 (baseline) and Days 1, 7, and 14
Placebo-corrected Change from Baseline in QRS Interval | Day -1 (baseline) and Days 1, 7, and 14
Number of Participants with Categorical Increases in QTcF from Baseline | Day -1 (baseline) and Days 1, 7, and 14
  Increases in absolute QTcF interval values from baseline >450 and ≤480 milliseconds (msec), >480 and ≤500 msec, or >500 msec, and changes from baseline of >30 and ≤60 msec, or >60 msec.
Number of Participants with Categorical Increases in PR Interval from Baseline | Day -1 (baseline) and Days 1, 7, and 14
  Increases in PR interval values from baseline >25% to a PR >200 msec.
Number of Participants with Categorical Increases in QRS Interval from Baseline | Day -1 (baseline) and Days 1, 7, and 14
  Increases in QRS interval from baseline >25% to a QRS >120 msec.
Number of Participants with Categorical Decreases in HR from Baseline | Day -1 (baseline) and Days 1, 7, and 14
  Decreases in HR from baseline >25% to a HR <50 beats per minute (bpm).
Change from Baseline in the Number of T-wave Morphology Findings | Day -1 (baseline) and Days 1, 7, and 14
Change from Baseline in the Number of U-waves | Day -1 (baseline) and Days 1, 7, and 14
Maximum Observed Plasma Concentration (Cmax) of Avacopan | Up to Day 14
Cmax of Avacopan Metabolite M1 | Up to Day 14
Time of Cmax (Tmax) of Avacopan | Up to Day 14
Tmax of Avacopan Metabolite M1 | Up to Day 14
Area Under the Plasma Concentration-time Curve (AUC) From Time 0 to 6 Hours (AUC0-6h) of Avacopan | Up to Hour 6 post-dose on Days 1, 7, and 14
AUC0-6h of Avacopan Metabolite M1 | Up to Hour 6 post-dose on Days 1, 7, and 14
AUC From Time 0 to 12 Hours (AUC0-12h) of Avacopan | Up to Hour 12 post-dose on Days 1, 7, and 14
AUC0-12h of Avacopan Metabolite M1 | Up to Hour 12 post-dose on Days 1, 7, and 14

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Derived] Miao S, Staehr P, Tai E, Darpo B, Xue H, Armas D, Webster K, Oberoi RK. A phase I thorough QT/QTc study evaluating therapeutic and supratherapeutic doses of avacopan in healthy participants. Clin Transl Sci. 2024 Jul;17(7):e13878. doi: 10.1111/cts.13878. PMID 38973157
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com